CLINICAL TRIAL: NCT03943797
Title: Cultivated Autologous Oral Mucosal Epithelial Transplantation for the Treatment of Ocular Surface Diseases: A Clinical Study
Brief Title: Cultivated Autologous Oral Mucosal Epithelial Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, David Hui-Kang Ma, Attending Physician, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101CONS12640; NCT02739113 (obsolete NCT alias)
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: Oral mucosal epithelial cells; Cornea; Amniotic membrane; Collagenase
MeSH Terms: conditions — Limbal Stem Cell Deficiency; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cultivated oral mucosal epithelial cell transplantation (Experimental): Cell therapy for treating severe limbal stem cell deficiency using cultivated autologous oral mucosal epithelial cells.
  Interventions: Biological: Cultivated oral mucosal epithelial cell transplantation

INTERVENTIONS:
Biological: Cultivated oral mucosal epithelial cell transplantation — Cultivated oral mucosal epithelial cell transplantation (COMET) will be used to treat severe limbal stem cell deficiency so as to restore the integrity of corneal surface

SUMMARY:
Earlier protocol for cultivated oral mucosal epithelial transplantation (COMET) requires trypsin/EDTA to isolate epithelial cells from tissue, and uses murine 3T3 cells as feeder cells, which results in biosafety concern. This study uses collagenase instead of trypsin/EDTA to isolate epithelial cells, and does not use 3T3 cells co-culture, so as to make an animal ingredient-free cell culture product. The purpose of the study is to evaluate the feasibility of the new protocol of COMET in clinical use.

DETAILED DESCRIPTION:
When corneal epithelial stem cells are destroyed by severe trauma such as burn or autoimmune diseases, poor regeneration of corneal epithelium, persistent inflammatory reaction, neovascular ingrowth, and conjunctivalization may ensue, and seriously reduce the vision. In treating the diseased eye, when the other eye is healthy, limbal tissue containing corneal epithelial stem cells can be harvested for direct tissue transplantation, or ex vivo cultivation and expansion for several days before transplantation.

For patients with bilaterally damaged eyes, rejection rate in non-HLA matched allograft limbal stem cell transplantation is very high, in addition, adverse reaction to long-term immunosuppressive therapy may be life-threatening. Therefore, in 2004 Japanese researchers first proposed a novel technique to treat ocular surface diseases using cultivated autologous oral mucosal epithelial transplantation (COMET). From 2006 to 2009, investigators have also conducted a Phase I clinical trial approved by Taiwan FDA. In that Phase I trial, investigators have demonstrated efficacy of such cell therapy in promoting wound healing in patients with severe ocular surface burns (Ma DHK et al. Eye 2009; 23: 1442- 1450). Investigators have also identify long-term persistence of transplanted oral mucosal epithelial cells in the cornea (Chen HCJ et al. IOVS 2009;50:4660-4668), justifying this innovative surgical procedure as an effective alternative treatment modality.

However, in previous protocol, animal products such as fetal calf serum and 3T3 cell culture were used, raising the biosafety concern. For this, recently investigators have developed an animal ingredient-free cell culture protocol, and our protocol can meet the GTP standards, and has obtained the accreditation by Taiwan FDA and affiliated institutes. Therefore, the focus of current Phase Ib trial is to confirm the feasibility and safety of following items:

1. To produce cell culture product not containing animal ingredient, so as to avoid zoonoses. The oral mucosal epithelial cells thus cultured are used for treating ocular surface diseases with limbal stem cell deficiency.
2. To reduce recurrence of corneal neovascularization after COMET, Bevacizumab (Avastin) is injected locally, so as to improve corneal transparency and visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Severe corneal epithelial deficiency
* Having favorable prognosis potential
* Normal of the intraocular pressure
* Normal of the light perception for the optic nerve
* No retinal diseases for the inflicted eyes
* No severe dry eye

Exclusion Criteria:

* Having unfavorable prognosis potential
* Severe systemic disorders
* Unable to use daily vision
* Mentally retarded to execute permit on surgery
* Pregnant woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of study specific AE | 12 months
  The tolerance and safety

CONTACTS AND LOCATIONS:
Overall Officials: David Hui-Kang Ma, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Core Laboratory for Cell Therapy, Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen HC, Chen HL, Lai JY, Chen CC, Tsai YJ, Kuo MT, Chu PH, Sun CC, Chen JK, Ma DH. Persistence of transplanted oral mucosal epithelial cells in human cornea. Invest Ophthalmol Vis Sci. 2009 Oct;50(10):4660-8. doi: 10.1167/iovs.09-3377. Epub 2009 May 20. PMID 19458337
- [Result] Chen HC, Yeh LK, Tsai YJ, Lai CH, Chen CC, Lai JY, Sun CC, Chang G, Hwang TL, Chen JK, Ma DH. Expression of angiogenesis-related factors in human corneas after cultivated oral mucosal epithelial transplantation. Invest Ophthalmol Vis Sci. 2012 Aug 17;53(9):5615-23. doi: 10.1167/iovs.11-9293. PMID 22850415
- [Result] Inatomi T, Nakamura T, Koizumi N, Sotozono C, Yokoi N, Kinoshita S. Midterm results on ocular surface reconstruction using cultivated autologous oral mucosal epithelial transplantation. Am J Ophthalmol. 2006 Feb;141(2):267-275. doi: 10.1016/j.ajo.2005.09.003. PMID 16458679
- [Result] Inatomi T, Nakamura T, Kojyo M, Koizumi N, Sotozono C, Kinoshita S. Ocular surface reconstruction with combination of cultivated autologous oral mucosal epithelial transplantation and penetrating keratoplasty. Am J Ophthalmol. 2006 Nov;142(5):757-64. doi: 10.1016/j.ajo.2006.06.004. Epub 2006 Sep 20. PMID 16989763
- [Result] Li W, Sabater AL, Chen YT, Hayashida Y, Chen SY, He H, Tseng SC. A novel method of isolation, preservation, and expansion of human corneal endothelial cells. Invest Ophthalmol Vis Sci. 2007 Feb;48(2):614-20. doi: 10.1167/iovs.06-1126. PMID 17251457
- [Result] Ma DH, Kuo MT, Tsai YJ, Chen HC, Chen XL, Wang SF, Li L, Hsiao CH, Lin KK. Transplantation of cultivated oral mucosal epithelial cells for severe corneal burn. Eye (Lond). 2009 Jun;23(6):1442-50. doi: 10.1038/eye.2009.60. Epub 2009 Apr 17. PMID 19373264
- [Result] Nakamura T, Inatomi T, Sotozono C, Amemiya T, Kanamura N, Kinoshita S. Transplantation of cultivated autologous oral mucosal epithelial cells in patients with severe ocular surface disorders. Br J Ophthalmol. 2004 Oct;88(10):1280-4. doi: 10.1136/bjo.2003.038497. PMID 15377551
- [Result] Nakamura T, Takeda K, Inatomi T, Sotozono C, Kinoshita S. Long-term results of autologous cultivated oral mucosal epithelial transplantation in the scar phase of severe ocular surface disorders. Br J Ophthalmol. 2011 Jul;95(7):942-6. doi: 10.1136/bjo.2010.188714. Epub 2010 Nov 19. PMID 21097786
- [Result] Petsoglou C, Balaggan KS, Dart JK, Bunce C, Xing W, Ali RR, Tuft SJ. Subconjunctival bevacizumab induces regression of corneal neovascularisation: a pilot randomised placebo-controlled double-masked trial. Br J Ophthalmol. 2013 Jan;97(1):28-32. doi: 10.1136/bjophthalmol-2012-302137. Epub 2012 Oct 20. PMID 23087419
- [Result] Satake Y, Higa K, Tsubota K, Shimazaki J. Long-term outcome of cultivated oral mucosal epithelial sheet transplantation in treatment of total limbal stem cell deficiency. Ophthalmology. 2011 Aug;118(8):1524-30. doi: 10.1016/j.ophtha.2011.01.039. Epub 2011 May 14. PMID 21571372
- [Result] Takeda K, Nakamura T, Inatomi T, Sotozono C, Watanabe A, Kinoshita S. Ocular surface reconstruction using the combination of autologous cultivated oral mucosal epithelial transplantation and eyelid surgery for severe ocular surface disease. Am J Ophthalmol. 2011 Aug;152(2):195-201.e1. doi: 10.1016/j.ajo.2011.01.046. Epub 2011 Jun 8. PMID 21652025
- [Result] Hsueh YJ, Huang SF, Lai JY, Ma SC, Chen HC, Wu SE, Wang TK, Sun CC, Ma KS, Chen JK, Lai CH, Ma DH. Preservation of epithelial progenitor cells from collagenase-digested oral mucosa during ex vivo cultivation. Sci Rep. 2016 Nov 8;6:36266. doi: 10.1038/srep36266. PMID 27824126
- [Derived] Ma DH, Hsueh YJ, Ma KS, Tsai YJ, Huang SF, Chen HC, Sun CC, Kuo MT, Chao AS, Lai JY. Long-term survival of cultivated oral mucosal epithelial cells in human cornea: generating cell sheets using an animal product-free culture protocol. Stem Cell Res Ther. 2021 Oct 7;12(1):524. doi: 10.1186/s13287-021-02564-7. PMID 34620226